CLINICAL TRIAL: NCT01724229
Title: An Open-Label Clinical Case Series to Demonstrate Efficacy of the Kendall Skin Wellness System
Brief Title: Clinical Case Series Evaluating Skin Wellness System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GM Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COV2012
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Moisture-associated Dermatitis; Fungal Infection in Perineal Area
Keywords: Incontinence-associated dermatitis; Skin care regimen for moisture-associated conditions; Perineal skin care; Fungal infection in perineal area

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment with OTC drug products (Other): * Body Wash & Shampoo applied directly to the skin or cloth; soiled area gently wiped clean. No rinsing necessary.
  * Moisture Barrier Cream: Once area cleansed and dried thoroughly, a thin coat is gently applied to the area of the skin exposed to moisture twice daily for two weeks or as directed by doctor.
  * 2-in-1 Cleanser: applied directly to the skin or a cloth and skin gently wiped clean. No rinsing necessary.
  * Antifungal Cream: Once reddened area cleansed and dried thoroughly a thin layer is applied over the affected area twice daily for two weeks or as directed by doctor.
  Interventions: Drug: Kendall Body Wash & Shampoo; Moisture Barrier Cream; 2-in-1 Cleanser; Antifungal Cream

INTERVENTIONS:
Drug: Kendall Body Wash & Shampoo; Moisture Barrier Cream; 2-in-1 Cleanser; Antifungal Cream

SUMMARY:
The purpose of this evaluation is to observe the performance of two (2) different skin care treatment protocols on the skin:

#1 Kendall™ Body Wash & Shampoo in combination with the Moisture Barrier Cream; or #2 Kendall™ 2-in-1 Cleanser in combination with the Anti-fungal Cream.

The scientific evidence supports using these types of skin care products to keep the skin healthy in the presence of moisture, urine, stool, or fungal infection. The cleansers are preferred over soap and water and can be applied on all areas of the skin. The Moisture Barrier Cream is formulated especially for skin exposed to moisture, urine, or stool. The Antifungal Cream is utilized for fungal infections associated with athlete's foot, jock itch, and ring worm to relieve itching, soreness, and irritation.

DETAILED DESCRIPTION:
The Kendall™ Body Wash & Shampoo is a no-rinse cleanser that gently removed dirt, urine, and stool while maintaining the natural pH of the skin (although it contains a shampoo component); it can be applied on all areas of the skin. Kendall™ Moisture Barrier Cream performs as a barrier to moisture and irritants when the natural barrier ability of the skin has been compromised.

Kendall™ 2-in-1 Cleanser is a no-rinse cleanser that gently removes dirt, urine, and stool and protects the skin from damage. Kendall™ Antifungal Cream is used on fungal infections to relieve itching and discomfort.

ELIGIBILITY:
Inclusion Criteria:

Adult subjects with any of the following indications:

* Erythema, maceration, or broken (denuded) skin from moisture, urinary or fecal incontinence
* Irritated, unbroken skin (perineal area)
* Fungal infection present in the perineal area

Exclusion Criteria:

* An existing pressure ulcer of any stage where the product will be applied
* Subjects not expected to survive the two week trial
* Subjects under age 18
* Subjects unable to provide informed consent (or whose designated power of attorney is unable to provide)
* Subjects with known sensitivity to any product preservative or other ingredient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
skin condition following treatment | 14 days
  Results of skin assessment will be documented using the IAD (Incontinence-Associated Dermatitis) Skin Condition Assessment Tool. Individual subscores will be added together to provide a ten-point scale for measurement of skin condition

CONTACTS AND LOCATIONS:
Overall Officials: Glenda J Motta, BSN, MPH, ET, Study Director — GM Associates Inc.
Locations (2):
- United States (2):
  - Villa Maria Care Center, Tucson, Arizona
  - Deer Meadows Retirement Community, Southampton, Pennsylvania

REFERENCES:
- [Background] Gray M, Beeckman D, Bliss DZ, Fader M, Logan S, Junkin J, Selekof J, Doughty D, Kurz P. Incontinence-associated dermatitis: a comprehensive review and update. J Wound Ostomy Continence Nurs. 2012 Jan-Feb;39(1):61-74. doi: 10.1097/WON.0b013e31823fe246. PMID 22193141
- [Background] Kennedy K, Leighton B, Lutz J. Cost-effectiveness evaluation of a new alchool-free, film-forming incontinence skin protectant. proceedings from the European Conference on Advances in Wound Management, Amsterdam, Oct. 1996